CLINICAL TRIAL: NCT04406311
Title: Italian Validation of the Low Anterior Resection Syndrome Score
Brief Title: Italian Validation of the LARS Score
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Carlo Ratto, Associate Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: LARS21052020
Record Dates: First submitted 2020-05-23; First posted 2020-05-28 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Rectal Cancer
Keywords: low anterior resection syndrome; Faecal incontinence; Quality of life; Soiling
MeSH Terms: conditions — Rectal Neoplasms; Low Anterior Resection Syndrome; Encopresis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BACKGROUND and RATIONALE Colorectal cancer, with 49,000 new diagnoses expected in 2019 (27,000 in men and 22,000 in women) represents, in Italy, the third neoplasm in men (14%) and the second in women (12%). Increasing attention has been recently paid to the outcomes of surgical treatment, in terms of patient's anorectal function and quality of life (QoL). Currently, the majority of patients affected by rectal carcinoma undergo a sphincter-sparing surgery, that is, a low anterior rectal resection (LAR).

It is known that about 50% - 90% of patients undergoing LAR will develop at least some degree of bowel dysfunction: for this reason, the definition of "anterior low rectal resection syndrome" (LARS) has been coined to describe this complex functional condition; the LARS usually includes incontinence to gas and/or liquid or solid stools, constipation, urgency, fragmentation and frequent bowel movements; a worsening of QoL has been also observed.

Due to the importance and high prevalence of this condition, but in the absence of a reliable tool for assessing its severity, the so-called "LARS score" has been introduced. The score has already been validated in several languages, even if this important tool has not been validated in Italian language.

AIMS of the STUDY The primary aim of this study will be the validation in Italian language of the LARS score in a population of Italian patients with a previous history of rectal cancer and treated by anterior rectal resection surgery. Moreover, the convergent and discriminatory validity, and the reliability of the score will be also assessed.

STUDY DESIGN The study will be a prospective observational study on patients affected by rectal cancer and treated by anterior rectal resection surgery with total or partial excision of the mesorectum (TME, total mesorectal excision, or PME, partial mesorectal excision) in the period January 2000 - April 2018. Any Unit of the Fondazione Policlinico Universitario "Agostino Gemelli" - IRCCS of Rome that deals with rectal cancer surgery could join the study.

METHODS The validated English version of the LARS questionnaire will be translated into Italian. The translation will be performed by two independent professional translators.

Based on previous validation studies conducted in other Countries, it has been calculated that the sample size will be 200 patients.

Patients will be assessed by administration of the LARS score questionnaire, of a single question on QoL, and of the EORTC-QLQ-C30 questionnaire.

Each Unit could choose to assess the patients in the preferred way (clinical follow-up visit, e-mail, ordinary mail); however, the method of administration of the questionnaire must be specified in the final communication of data to the coordinating Group. Each Unit joining the Study will be provided with an Excel data collection sheet which must then be completed.

A descriptive analysis of the data will be conducted, and the convergent validity, that is the concordance between the LARS score and the QoL, will be investigated. In addition, discriminatory validity, i.e. the ability of the LARS score to distinguish between subgroups of patients, which usually differ in the LARS score, will be assessed. Finally, the test-retest reliability of the LARS score will be examined, so all patients will receive a second LARS questionnaire 1-2 weeks after completing the first and the results of the two tests will be compared.

DETAILED DESCRIPTION:
1. BACKGROUND and RATIONALE Colorectal cancer, with 49,000 new diagnoses expected in 2019 (27,000 in men and 22,000 in women) represents, in Italy, the third neoplasm in men (14%) and the second in women (12%). Among colorectal tumors, the rectum represents the site most frequently involved (about 35%).

   Thanks to an earlier diagnosis and to the greater effectiveness of an implemented multidisciplinary treatment, the locoregional control and the patients' overall survival significantly improved over the last decades.

   Increasing attention has been recently paid to the outcomes of surgical treatment, in terms of patient's anorectal function and quality of life (QoL). Currently, the majority of patients affected by rectal carcinoma undergo a sphincter-sparing surgery, that is, a low anterior rectal resection (LAR), therefore avoiding a permanent colostomy.

   It is known that about 50% - 90% of patients undergoing LAR will have at least some degree of bowel dysfunction: for this reason, the definition of "anterior low rectal resection syndrome" (LARS) has been coined to describe this complex functional condition. The main symptoms included in this syndrome are: incontinence to gas and/or liquid or solid stools, constipation, urgency, fragmentation and frequent bowel movements. In addition, a worsening of QoL has been observed in patients with severe LARS symptoms.

   Due to the importance and high prevalence of this condition, in order to identify a reliable tool for assessing its severity, the so-called "LARS score" has been introduced. The score has already been validated in several languages, including English, Chinese, Lithuanian, Swedish, Spanish, German, Danish (as consolidated international validation), and finally Dutch.

   However, this important tool has not been validated in Italian language.
2. AIMS The primary aim of this study will be the validation in Italian language of the LARS score in a population of Italian patients with a previous history of rectal cancer, and treated by anterior rectal resection surgery. Moreover, the study will give the possibility to investigate the convergent and discriminatory validity, and to re-test the reliability of the score.
3. STUDY DESIGN The study will be a prospective observational study on patients affected by rectal cancer, and treated by anterior rectal resection surgery with total or partial excision of the mesorectum (TME, total mesorectal excision, or PME, partial mesorectal excision) in the period January 2000 - April 2018. Any Surgical Unit of the Fondazione Policlinico Universitario "Agostino Gemelli" - IRCCS of Rome that deals with rectal cancer surgery could join the study. Each Unit will identify a Study Manager, and possibly a collaborator.
4. METHODS

   The study will provide different phases:
   * TRANSLATION OF THE QUESTIONNAIRE The validated English version of the LARS questionnaire will be translated into Italian. The translation will be performed by two independent professional translators. Translators will discuss any discrepancies between their translations until an agreed version is reached. A third native English translator will translate the Italian version into English. Subsequently, the two English versions (the initial one and the new one) will be compared and the final version in Italian will be elaborated.
   * CONVERGENT VALIDITY To study the "convergent validity", the LARS score will be correlated with the single QoL question and with the EORTC-QLQ-C30 questionnaire, in order to test how the LARS score correlates with the QoL.
   * DIVERGENT VALIDITY To study discriminative validity, we will evaluate the ability of the LARS score to identify different patient subgroups, which generally differ in the LARS score. Similar to previous validation studies, the clinically relevant subgroups will be based on: preoperative radiotherapy, type of surgery (TME / PME), age (cut-off at 69 years).
   * TEST- RETEST RELIABILITY Test-retest reliability is one of the key measures of all health measures. To examine the test-retest reliability of the LARS score, all patients will receive a second LARS questionnaire 1-2 weeks after completing the first one, and will be invited to reply to the questionnaire again.

   Each Unit could choose to assess the patients in the preferred way (clinical follow-up visit, e-mail, ordinary mail); however, the method of administration of the questionnaire must be specified in the final communication of data to the coordinating Group.

   Each Unit will be responsible for the truthfulness of the data collected and provided.
5. DATA COLLECTION

   Each Unit joining the Study will be provided with an Excel data collection sheet which must then be completed. The collection of data and their transmission to the Study Coordinator Group must occur within 3 months from the beginning of the Study. For each patient we ask to provide:
   * 2 LARS questionnaires, administered 1-2 weeks apart;
   * 1 EORTC-QLQ-C30 questionnaire;
   * 1 single QoL question.
6. STATISTICAL ANALYSIS and DATA EVALUATION The quality control of the collected data and the statistical analysis of the results will be conducted by a specialist in Medical Statistics, who will be guaranteed co-authorship in the scientific publications derived from the study. No financial compensation will be provided for this activity.

   Concerning the "convergent validity", the correspondence between the QoL categories (no impact, minor or major impact of intestinal function on QoL) and the three LARS scoring categories will be assessed. The correspondence between these two measures will be considered perfect when: patients have not reported LARS and any impact on QoL; patients have reported minor LARS and a minor impact on QoL; in case of major LARS and major impact on QoL. Correspondence will be defined as moderate in case of a difference in one category, for example no LARS but a minor impact on QoL. In case of difference in two categories, the two measures will be considered not corresponding at all.

   LARS score data will be presented as median (with interquartile range) and the differences will be tested by the Kruskal-Wallis test. The same test will be used to test the null hypothesis in the study of the association between the LARS score and the five functional scales and the global QoL scale of the EORTC-QLQ-C30 questionnaire. Wilcoxon's rank test will be applied to investigate the "discriminatory validity".

   The correspondence between the two tests to measure the reliability of the LARS score will be presented as proportions with 95% confidence intervals (95% CI). A Bland-Altman diagram will be calculated with 95% agreement limits and intraclass correlation (ICC). An ICC lower than 0.50 will indicate poor reliability, an ICC between 0.50 and 0.75 will reflect moderate reliability, between 0.75-0.90 good reliability and an ICC greater than 0.90 will indicate excellent reliability.
7. PUBLICATION POLICY and AUTHORSHIP The results of the study will be the subject of a group publication. The co-authorship of the manager and a collaborator will be guaranteed to each Unit participating in the study. The first, second and last Author of the publication will be respectively the principal investigator and the two collaborators (junior and senior) of the promoter / coordinator Center.

ELIGIBILITY:
Inclusion Criteria:

* rectal neoplasia (between 0 and 15 cm from the anal verge);
* anterior rectal resection surgery with total or partial mesorectal excision (TME or PME) in the period January 2000 - April 2018;
* if a stoma had been created, intestinal continuity must have been restored for at least 24 months (by April 2018);

Exclusion Criteria:

* dementia;
* metastatic or recurrent disease;
* other intestinal diseases (including Crohn's disease, ulcerative colitis);
* patients with a stoma or with intestinal continuity restored for less than 24 months;
* patients with problems of understanding the Italian language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a previous diagnosis of rectal neoplasia, who underwent anterior rectal resection surgery with total or partial mesorectal excision (TME or PME) at "Fondazione Policlinico Agostino Gemelli IRCCS" in Rome
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Lars score | June 2020- August 2020
  The LARS score, originally developed in Denmark, aims to assess the intestinal dysfunction in a population of rectal cancer patients. The sum of the scores of the five subscales allows to calculate a total score ranging from 0 to 42 points. So, the total score is classified into three groups: 0-20 points: no LARS; 21-29 points: minor LARS; 30-42 points: major LARS.

SECONDARY OUTCOMES:
EORTC-QLQ-C30 questionnaire | June 2020- August 2020
  The EORTC-QLQ-C30 questionnaire is a validated and specific tool to evaluate the QoL of cancer patients. It consists of 30 questions that provide a global QoL scale, five functional scales (i.e. physical, role-playing, emotional, cognitive, social), three symptom scales (fatigue, nausea and vomiting, pain) and six individual factors (dyspnea, insomnia, loss of appetite, constipation, diarrhea, financial difficulties). The scores of each scale are calculated in a score ranging from 0 to 100. For the purpose of this study, only the functional scales and the global QoL scale will be used. A high score on a functional scale represents a good level of function.
Single question on QoL | June 2020- August 2020
  A single question on QoL will be added to the LARS score for the purpose of investigating convergent validity. The question is: "Overall, how does bowel function affect your quality of life?"; it will be possible to give only one of the following answers: "not at all", "a little", "enough", "a lot". This question had previously been used for the development and validation of the LARS score in other countries. The score ranges from 0 to 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico universitario Agostino Gemelli, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Emmertsen KJ, Laurberg S. Bowel dysfunction after treatment for rectal cancer. Acta Oncol. 2008;47(6):994-1003. doi: 10.1080/02841860802195251. PMID 18607875
- [Background] Bryant CL, Lunniss PJ, Knowles CH, Thaha MA, Chan CL. Anterior resection syndrome. Lancet Oncol. 2012 Sep;13(9):e403-8. doi: 10.1016/S1470-2045(12)70236-X. PMID 22935240
- [Background] Juul T, Ahlberg M, Biondo S, Espin E, Jimenez LM, Matzel KE, Palmer GJ, Sauermann A, Trenti L, Zhang W, Laurberg S, Christensen P. Low anterior resection syndrome and quality of life: an international multicenter study. Dis Colon Rectum. 2014 May;57(5):585-91. doi: 10.1097/DCR.0000000000000116. PMID 24819098
- [Background] Emmertsen KJ, Laurberg S. Low anterior resection syndrome score: development and validation of a symptom-based scoring system for bowel dysfunction after low anterior resection for rectal cancer. Ann Surg. 2012 May;255(5):922-8. doi: 10.1097/SLA.0b013e31824f1c21. PMID 22504191
- [Background] Juul T, Battersby NJ, Christensen P, Janjua AZ, Branagan G, Laurberg S, Emmertsen KJ, Moran B; UK LARS Study Group. Validation of the English translation of the low anterior resection syndrome score. Colorectal Dis. 2015 Oct;17(10):908-16. doi: 10.1111/codi.12952. PMID 25807963
- [Background] Hou XT, Pang D, Lu Q, Yang P, Jin SL, Zhou YJ, Tian SH. Validation of the Chinese version of the low anterior resection syndrome score for measuring bowel dysfunction after sphincter-preserving surgery among rectal cancer patients. Eur J Oncol Nurs. 2015 Oct;19(5):495-501. doi: 10.1016/j.ejon.2015.02.009. Epub 2015 Mar 23. PMID 25813530
- [Background] Samalavicius NE, Dulskas A, Lasinskas M, Smailyte G. Validity and reliability of a Lithuanian version of low anterior resection syndrome score. Tech Coloproctol. 2016 Apr;20(4):215-20. doi: 10.1007/s10151-015-1424-0. Epub 2016 Jan 12. PMID 26754654
- [Background] Juul T, Ahlberg M, Biondo S, Emmertsen KJ, Espin E, Jimenez LM, Matzel KE, Palmer G, Sauermann A, Trenti L, Zhang W, Laurberg S, Christensen P. International validation of the low anterior resection syndrome score. Ann Surg. 2014 Apr;259(4):728-34. doi: 10.1097/SLA.0b013e31828fac0b. PMID 23598379
- [Background] Hupkens BJP, Breukink SO, Olde Reuver Of Briel C, Tanis PJ, de Noo ME, van Duijvendijk P, van Westreenen HL, Dekker JWT, Chen TYT, Juul T. Dutch validation of the low anterior resection syndrome score. Colorectal Dis. 2018 Oct;20(10):881-887. doi: 10.1111/codi.14228. Epub 2018 May 16. PMID 29679514
- [Background] Aaronson NK, Ahmedzai S, Bergman B, Bullinger M, Cull A, Duez NJ, Filiberti A, Flechtner H, Fleishman SB, de Haes JC, et al. The European Organization for Research and Treatment of Cancer QLQ-C30: a quality-of-life instrument for use in international clinical trials in oncology. J Natl Cancer Inst. 1993 Mar 3;85(5):365-76. doi: 10.1093/jnci/85.5.365. PMID 8433390
- [Background] Fayers PM. Interpreting quality of life data: population-based reference data for the EORTC QLQ-C30. Eur J Cancer. 2001 Jul;37(11):1331-4. doi: 10.1016/s0959-8049(01)00127-7. No abstract available. PMID 11435060
- [Background] Klee M, Groenvold M, Machin D. Using data from studies of health-related quality of life to describe clinical issues examples from a longitudinal study of patients with advanced stages of cervical cancer. Qual Life Res. 1999 Dec;8(8):733-42. doi: 10.1023/a:1008903818379. PMID 10855347
- [Background] Bregendahl S, Emmertsen KJ, Lous J, Laurberg S. Bowel dysfunction after low anterior resection with and without neoadjuvant therapy for rectal cancer: a population-based cross-sectional study. Colorectal Dis. 2013 Sep;15(9):1130-9. doi: 10.1111/codi.12244. PMID 23581977
- [Background] Polit DF. Getting serious about test-retest reliability: a critique of retest research and some recommendations. Qual Life Res. 2014 Aug;23(6):1713-20. doi: 10.1007/s11136-014-0632-9. Epub 2014 Feb 7. PMID 24504622
- [Background] Landis JR, Koch GG. The measurement of observer agreement for categorical data. Biometrics. 1977 Mar;33(1):159-74. PMID 843571
- [Derived] De Simone V, Litta F, Persiani R, Rizzo G, Sofo L, Menghi R, Santullo F, Biondi A, Coco C, Sacchetti F, Longo F, Attalla El Halabieh M, Moroni R, Ratto C. Effectiveness and Validation of the Italian Translation of the Low Anterior Resection Syndrome Score in an Italian High-Volume University Hospital. Front Surg. 2022 Jun 20;9:917224. doi: 10.3389/fsurg.2022.917224. eCollection 2022. PMID 35795231
- See also: Related Info — http://www.aiom.it/wp-content/uploads/2019/09/2019_Numeri_Cancro-operatori-web.pdf